CLINICAL TRIAL: NCT05419999
Title: Safety, Feasibility, and Benefits of Transcranial Direct Current Stimulation (tDCS) in Human Subjects With Posttraumatic Stress Disorder (PTSD) Receiving an Exposure-based, Behavioral Therapy
Brief Title: Transcranial Direct Current Stimulation (tDCS) in Human Subjects With PTSD Receiving an Exposure-based, Behavioral Therapy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: The University of Texas Health Science Center at San Antonio (Other)
Responsible Party: Principal Investigator, Casey Straud, Associate Professor, The University of Texas Health Science Center at San Antonio
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: HSC20220158H
Record Dates: First submitted 2022-06-10; First posted 2022-06-15 (Actual); Results first posted 2025-05-29 (Actual); Last update posted 2025-05-29 (Actual); Status verified 2025-05

CONDITIONS: Post Traumatic Stress Disorder
Keywords: Brain stimulation
MeSH Terms: conditions — Stress Disorders, Post-Traumatic

STUDY DESIGN:
Intervention Model Description: Early phase II, two-arm, partially double-blind pilot research clinical trial
Who Masked: Participant
Masking Description: Subjects will be blinded to whether they receive actual tDCS or sham treatment. All study team members will also be blinded to randomization, with the exception of the study team coordinator who will allocate device codes. This will allow for the blind to be broken in case of an emergency or serious adverse event.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (2):
- tDCS plus WET (Experimental): Subjects will receive transcranial direct current stimulation (tDCS) plus written exposure therapy (WET)
  Interventions: Device: Soterix 1x1 tDCS mini CT; Behavioral: Written Exposure Therapy (WET)
- Sham plus WET (Sham Comparator): Subjects will receive sham transcranial direct current stimulation (tDCS) treatment plus written exposure therapy (WET)
  Interventions: Other: Sham Soterix 1x1 tDCS Mini CT; Behavioral: Written Exposure Therapy (WET)

INTERVENTIONS:
Device: Soterix 1x1 tDCS mini CT — During stimulation, a current flows between the electrodes passing through the brain to complete the circuit. tDCS is hypothesized to modulate intrinsic neuronal activity by enhancing neuronal resting potential, or altering the likelihood that a neuron will (or will not) depolarize.
  Other Names: Transcranial Direct Current Stimulator
  Arms: tDCS plus WET
Other: Sham Soterix 1x1 tDCS Mini CT — Sham setting is used on the Soterix transcranial electrical stimulator
  Other Names: Sham Transcranial Direct Current Stimulator
  Arms: Sham plus WET
Behavioral: Written Exposure Therapy (WET) — An exposure-based, behavioral psychotherapy for PTSD.

SUMMARY:
The primary objective of this study is to evaluate the safety, feasibility, and psychological and physiological treatment benefits of transcranial direct current stimulation (tDCS), a noninvasive brain stimulation technique, when delivered in combination with Written Exposure Therapy (WET), for posttraumatic stress disorder posttraumatic stress disorder (PTSD).

DETAILED DESCRIPTION:
While the potential for non-invasive brain stimulation is exciting, research is needed to determine the safety, feasibility, and benefits of non-invasive brain stimulation in human subjects with PTSD. Towards this end, the study team will conduct a single-blind randomized controlled pilot study of transcranial direct current stimulation (tDCS) vs. a sham condition in a sample of 40 adults with PTSD receiving 5 weekly sessions of Written Exposure Therapy (WET), an exposure-based, behavioral psychotherapy for PTSD.

ELIGIBILITY:
Inclusion Criteria:

1. Individuals between the ages of 18 and 65 years old at time of screening.
2. PTSD diagnosis as assessed by the Clinician-Administered Posttraumatic Stress Scale (CAPS-5)
3. Able to write, read, and speak English

Exclusion Criteria:

1. History of epilepsy or seizures.
2. History of significant intracranial pathology (e.g., severe traumatic brain injury) or neurological disorder (e.g., Stroke, Multiple Sclerosis, Amyotrophic Lateral Sclerosis, Alzheimer's, Dementia, Parkinson's, and/or Huntington's).
3. History of skin condition (e.g., eczema, psoriasis) where electrodes will be applied.
4. Electronic implants in the body that could be susceptible to electrical current (e.g., cardiac pacemaker, cochlear implants, medical pump).
5. Metallic objects other than dental appliances/fillings near the site of stimulation
6. Current manic episode or psychotic symptoms requiring immediate stabilization or hospitalization (as determined by clinical judgement).
7. Current moderate or severe substance use disorder.
8. Suicidality and/or psychiatric risk requiring immediate intervention or a higher level of care than can be provided by the study treatment.
9. Change in anticonvulsive or benzodiazepine medication regimen in the past month.
10. History of adverse effects to previous tDCS or other brain stimulation technique.
11. Concurrent engagement in another brain simulation technique or trauma-related psychotherapy for PTSD.
12. Currently pregnant or breastfeeding.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 25 (Actual)
Dates: Start 2023-01-09 (Actual); Primary Completion 2024-04-25 (Actual); Study Completion 2024-04-25 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Casey Straud, PsyD, Principal Investigator — University of Texas Health Science Center San Antonio
Locations (1):
- The University of Texas Health Science Center at San Antonio, San Antonio, Texas, United States

IPD SHARING:
Plan to Share IPD: Yes
At the conclusion of this study, participants who signed the consent to have their data placed in the STRONG STAR Repository will be maintained under the UTHSCSA IRB-approved Repository protocol. For participants who decline participation in the STRONG STAR Repository, at the conclusion of the study their data will be de-identified and the data maintained in the Repository without identifiers. The IRB approved STRONG STAR Repository is a large comprehensive database of information, biological specimens and neuroimages related to the identification, assessment, and treatment of posttraumatic stress disorder (PTSD), insomnia, pain, and related behavioral health conditions. No biospecimen data is being collected in this study.
Supporting Information: Study Protocol, SAP
Time Frame: Anticipated study duration is 24 months to obtaining, cleaning and analysis of the data.

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | tDCS Plus WET | Sham Plus WET
Started | 12 | 13
Completed | 12 | 12
Not Completed | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | tDCS Plus WET | Sham Plus WET | Total
Number analyzed (Participants) | 12 | 13 | 25
Age, Continuous [Mean (Standard Deviation); unit: years] | 42.67 (6.54) | 39.00 (9.75) | 40.76 (8.40)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5 | 4 | 9
  Male | 7 | 9 | 16
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1 | 0 | 1
  Asian | 1 | 0 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 1 | 2 | 3
  White | 9 | 11 | 20
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 12 | 13 | 25

OUTCOME MEASURES:

1. Primary Outcome: Posttraumatic Stress Disorder Checklist (PCL-5)
Description: The PCL-5 is a 20-item self-report measure update of the PCL designed to assess PTSD symptoms as defined by the DSM-5. The PCL-5 is currently available and has been shown to have good psychometric properties. The PCL-5 evaluates how much participants have been bothered by PTSD symptoms in the past week (for all assessments during treatment) or the past two weeks (all other assessment time points) as a result of a specific life event. Each item of the PCL-5 is scored on a five-point scale ranging from 0 "not at all") to 4 ("extremely). This measure will be administered at the baseline assessment, prior to each therapy session, and the one-month follow-up assessment. The potential scores range from 0-80, with a lower score indicating less symptoms of PTSD.
Time Frame: Baseline to 9 weeks (one month post study treatment)
Measure: Mean (Standard Error); unit: score on a scale
Arm/Group | tDCS Plus WET | Sham Plus WET
Number analyzed (Participants) | 12 | 13
score on a scale
  BASELINE | 44.30 (3.74) | 43.38 (3.56)
  9 WEEKS | 22.51 (3.98) | 25.11 (3.78)

2. Primary Outcome: Number of Subjects That Completed All 5 WET Sessions
Description: Tracking feasibility through number of subjects that complete all written exposure therapy
Time Frame: 5 weeks
Measure: Count of Participants; unit: Participants
Arm/Group | tDCS Plus WET | Sham Plus WET
Number analyzed (Participants) | 12 | 13
Participants | 12 | 12

3. Secondary Outcome: Clinician Administer PTSD Scale-5 (CAPS-5)
Description: The CAPS-5 is structured interview that assesses the DSM-5 criteria for PTSD. Each item is rated on a severity scale ranging from 0 (Absent) to 4 (Extreme/incapacitating) and combines information about frequency and intensity for each of the 20 symptoms. Additional items that are not included in the total score evaluate overall symptom duration, distress, impairment, dissociative symptoms, and global ratings by the interviewer. Scores range from 0-80, with lower scores indicating less PTSD severity.
Time Frame: Baseline to 9 weeks (one month post study treatment)
Measure: Mean (Standard Error); unit: score on a scale
Arm/Group | tDCS Plus WET | Sham Plus WET
Number analyzed (Participants) | 12 | 13
score on a scale
  BASELINE | 35.95 (2.01) | 35.08 (1.93)
  9 WEEKS | 14.65 (2.31) | 15.89 (2.09)

4. Secondary Outcome: Patient Health Questionnaire-9 (PHQ)
Description: The PHQ-9 is a widely used and well-validated instrument for measuring the severity of depressive symptoms. It consists of 9 items that assess both affective and somatic symptoms related to depression and depressive disorders. Respondents rate the frequency with which they have been bothered by depressive symptoms within the past two weeks on a scale ranging from 0 ("not at all") to 3 ("nearly every day"). Scores range from 0-27, with lower scores indicating less depression severity.
Time Frame: Baseline to 9 weeks (one month post study treatment)
Measure: Mean (Standard Error); unit: score on a scale
Arm/Group | tDCS Plus WET | Sham Plus WET
Number analyzed (Participants) | 12 | 13
score on a scale
  BASELINE | 15.58 (1.82) | 15.54 (1.75)
  9 WEEKS | 11.00 (2.07) | 10.66 (1.88)

5. Secondary Outcome: Generalize Anxiety Disorder-7 (GAD)
Description: The GAD-7will be used to assess generalized anxiety symptomology. This is a 7-item measure that asks participants to rate the frequency with which they have been bothered by anxiety symptoms within the past two weeks on a scale ranging from 0 ("not at all") to 3 ("nearly every day"). Scores range from 0-21, with lower scores indicating less anxiety severity.
Time Frame: Baseline to 9 weeks (one month post study treatment)
Measure: Mean (Standard Error); unit: score on a scale
Arm/Group | tDCS Plus WET | Sham Plus WET
Number analyzed (Participants) | 12 | 13
score on a scale
  BASELINE | 15.00 (1.61) | 15.39 (1.55)
  9 WEEKS | 10.30 (1.76) | 9.74 (1.60)

ADVERSE EVENTS:
Time Frame: Adverse events were assessed at every visit following the baseline assessment. Participants were assessed for AEs at sessions 1 through 5 and at the 1-month follow-up (9-weeks)
Description: At each session, participants are asked "Have you experienced any changes for the worse since your last visit?" All reported events were documented by the research team member. Participants were also asked about the temporal nature (start/stop date), severity, impact on functioning, and whether the event is study-related or attributable to something else.
Arm/Group | tDCS Plus WET | Sham Plus WET
All-Cause Mortality (participants affected / at risk) | 0/12 | 0/13
Serious Adverse Events (participants affected / at risk) | 0/12 | 0/13
Other Adverse Events (participants affected / at risk) | 10/12 | 11/13
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | tDCS Plus WET (N=12) | Sham Plus WET (N=13)
Emotional Distress (Psychiatric disorders) | 5 (7) | 5 (9)
Pain (Musculoskeletal and connective tissue disorders) | 4 (4) | 3 (3) — Pain in area other than stimulation site (foot, jaw, muscle, neck, throat)
Irritability (Psychiatric disorders) | 4 (4) | 2 (2)
Anxiety (Psychiatric disorders) | 6 (7) | 2 (2)
Reexperiencing (Psychiatric disorders) | 3 (3) | 2 (2)
Sleep Disturbance (Psychiatric disorders) | 4 (6) | 3 (3)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2024-05-14): https://cdn.clinicaltrials.gov/large-docs/99/NCT05419999/Prot_SAP_000.pdf
  • Informed Consent Form (2024-05-14): https://cdn.clinicaltrials.gov/large-docs/99/NCT05419999/ICF_001.pdf